CLINICAL TRIAL: NCT01300845
Title: Prospective, Randomized, Multi-center Trial Aiming at Assessing the Effect of Humidification on the Comfort of the Patient Receiving an Oxygen Therapy.
Brief Title: Trial Aiming at Assessing the Effect of Humidification on the Comfort of the Patient Receiving an Oxygen Therapy
Acronym: OXYREA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHRI 2010-02
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-02

CONDITIONS: Oxygen Inhalation Therapy
Keywords: Oxygen mask; Oxygen cannula; Humidification; Oxygen therapy; Intensive Care Unit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Humidification (Active Comparator)
  Interventions: Procedure: Humidification
- No Humidification (Experimental)
  Interventions: Procedure: No Humidification

INTERVENTIONS:
Procedure: Humidification — From randomization, oxygen therapy is humidified
  Arms: Humidification
Procedure: No Humidification — oxygen therapy is never humidified
  Arms: No Humidification

SUMMARY:
In France, the most used humidifying system during oxygen therapy is a non heated device with weak efficiency and non-proven clinical benefits. This study aims to assess the lack of benefits of non-heated humidification compared to no humidification, as regards to the comfort of the patient receiving oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Admission in Intensive Care Unit
* Oxygen therapy started for less than two hours in ICU

Exclusion Criteria:

* Age under 18
* Pregnancy
* Participation in other trials with the same endpoints
* absence of registration in french health care system
* patient protected by law
* tracheotomised or intubated patient
* Patient with non invasive ventilation
* Oxygen therapy started for more than two hours in ICU
* moribund

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2011-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
A score of comfort assessed with a detailed and specific questionnaire | This score is assessed between the sixth and the eighth hour after randomization
  This score is built from answers brought in a questionnaire including 15 items. Each item can be rated from 0 to 10, allowing to increment a score on 150 points.

SECONDARY OUTCOMES:
The specific scores of comfort for each items | Hour 6-8
Observance level for oxygen therapy | Hour 6-8
Percentage of patients requiring a fibroscopic aspirations during their stay in intensive care unit or USC within the limits of 28 days. | Department discharge limited by day 28
Percentage of patients requiring an intubation during their stay in intensive care unit or USC within the limits of 28 days. | Department discharge limited by day 28
Percentage of patients who had an ear, nose and throat infections during their stay in intensive care unit or USC within the limits of 28 days. | Department discharge limited by day 28
The patients who had a lesion of corneas during their stay in intensive care unit or USC within the limits of 28 days | Department discharge limited by day 28
The length of stay in intensive care unit or USC | Department discharge limited by day 28
mortality in intensive care unit or USC during ongoing stay within the limits of 28 days. | Department discharge limited by day 28

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Angers, France